CLINICAL TRIAL: NCT00597207
Title: A Randomized Controlled Study Comparing Autopulse To Manual CPR In A CPR-First Protocol For Out-Of-Hospital Cardiac Arrest
Brief Title: Circulation Improving Resuscitation Care (CIRC)
Acronym: CIRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Collaborators: Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zoll-0100
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: CPR; mechanical; manual; outcome; survival; quality
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mechanical CPR with AutoPulse
  Interventions: Device: AutoPulse
- 2 (Other): Manual CPR
  Interventions: Other: Manual

INTERVENTIONS:
Device: AutoPulse — Mechanical device that provides chest compression
  Arms: 1
Other: Manual — Manual chest compression
  Arms: 2

SUMMARY:
During resuscitation of out of hospital cardiac arrest patients the use of a mechanical chest compression device Autopulse will improve survival compared to manual compressions.

DETAILED DESCRIPTION:
Sudden out-of-hospital cardiac arrest (OOH-CA) remains a significant cause of death, in spite of recent declines in overall mortality from cardiovascular disease. Several studies document sub optimal quality of manual chest compressions and this may influence outcome. However, studies comparing manual and mechanical chest compressions have resulted in conflicted results. The investigators think this may be based on methodology and design issues of the trials as much as not focusing on training and experience in operating a mechanical device clinically. Therefore the investigators will focus on these issues and implement three phases in the study (In field training, Run In phase, and Study phase). The investigators will also focus on early use of mechanical CPR after arrival at patient side and randomization at arrival. In order to achieve this the investigators will follow the Norwegian CPR Guidelines with 3 min CPR before defibrillation and the 3 min algorithm. Quality of CPR will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patents aged 18 years (or local age of consent) or more who suffer non-traumatic arrest of presumed cardiac etiology in an out-of-hospital setting and who do not meet any of the exclusion criteria below.

Exclusion Criteria:

* Traumatic arrest (blunt, penetrating, burns)
* Arrest due to exsanguinations, strangulation, smoke inhalation, drug overdose, electrocution, hanging, drowning.
* Known or clinically apparent pregnancy
* Do Not Attempt to Resuscitate (DNAR) orders
* Apparent patient weight more than 225 kg (500 lbs)
* Wards of the state
* Prisoner
* CPR device other than AutoPulse
* Patients who are reached after 16 minutes after the time of emergency call (911). This exclusion is determined at the time of CRF abstraction, not during treatment of the patient.

  * If patient is unaccompanied, or accompanied by a person or persons unfamiliar with their his-tory, determination of these exclusion criteria will, perforce, be left to the best estimation of the rescue personnel. At no time, should an attempt to determine these criteria be allowed to delay the administration of life-saving treatment.

    * These criteria will be determined in the best estimation of the rescue personnel, or if the AutoPulse signals that the patient is outside the parameters for AutoPulse deployment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4231 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, Principal Investigator — Ullevaal University Hospital; David Persse, MD, Principal Investigator — Houston Fire
Locations (5):
- United States (3):
  - Hillsborough Fire Rescue, Tampa, Florida
  - Houston Fire, Houston, Texas
  - Gold Cross EMS, Menasha, Wisconsin
- Vienna EMS, Vienna, Austria
- Nijmegen EMS, Nijmegen, Netherlands

REFERENCES:
- [Derived] Olsen JA, Brunborg C, Steinberg M, Persse D, Sterz F, Lozano M Jr, Westfall M, van Grunsven PM, Lerner EB, Wik L. Survival to hospital discharge with biphasic fixed 360 joules versus 200 escalating to 360 joules defibrillation strategies in out-of-hospital cardiac arrest of presumed cardiac etiology. Resuscitation. 2019 Mar;136:112-118. doi: 10.1016/j.resuscitation.2019.01.020. Epub 2019 Jan 29. PMID 30708074
- [Derived] Wik L, Olsen JA, Persse D, Sterz F, Lozano M Jr, Brouwer MA, Westfall M, Souders CM, Travis DT, Herken UR, Lerner EB. Why do some studies find that CPR fraction is not a predictor of survival? Resuscitation. 2016 Jul;104:59-62. doi: 10.1016/j.resuscitation.2016.04.013. Epub 2016 May 4. PMID 27155547
- [Derived] Steinberg MT, Olsen JA, Brunborg C, Persse D, Sterz F, Lozano M Jr, Brouwer MA, Westfall M, Souders CM, van Grunsven PM, Travis DT, Lerner EB, Wik L. Minimizing pre-shock chest compression pauses in a cardiopulmonary resuscitation cycle by performing an earlier rhythm analysis. Resuscitation. 2015 Feb;87:33-7. doi: 10.1016/j.resuscitation.2014.11.012. Epub 2014 Nov 21. PMID 25461493
- [Derived] Wik L, Olsen JA, Persse D, Sterz F, Lozano M Jr, Brouwer MA, Westfall M, Souders CM, Malzer R, van Grunsven PM, Travis DT, Whitehead A, Herken UR, Lerner EB. Manual vs. integrated automatic load-distributing band CPR with equal survival after out of hospital cardiac arrest. The randomized CIRC trial. Resuscitation. 2014 Jun;85(6):741-8. doi: 10.1016/j.resuscitation.2014.03.005. Epub 2014 Mar 15. PMID 24642406
- [Derived] Lerner EB, Persse D, Souders CM, Sterz F, Malzer R, Lozano M Jr, Westfall M, Brouwer MA, van Grunsven PM, Whitehead A, Olsen JA, Herken UR, Wik L. Design of the Circulation Improving Resuscitation Care (CIRC) Trial: a new state of the art design for out-of-hospital cardiac arrest research. Resuscitation. 2011 Mar;82(3):294-9. doi: 10.1016/j.resuscitation.2010.11.013. Epub 2010 Dec 31. PMID 21196070

RESULTS

PARTICIPANT FLOW:
Groups:
- iA-CPR: Integrated Mechanical CPR with AutoPulse All subjects initially receive manual chest compressions. After randomization, subjects randomized to iA-CPR are moved to the device once it is ready and from thereon receive mechanical chest compressions.
  AutoPulse: Mechanical device that provides chest compression
- M-CPR: Manual CPR All subjects initially receive manual chest compressions. After randomization, subjects randomized to M-CPR continue to receive manual chest compressions.
  Manual: Manual chest compression
Period: Overall Study
Arm/Group | iA-CPR | M-CPR
Started | 2099 | 2132
Completed | 2094 | 2125
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iA-CPR | M-CPR | Total
Number analyzed (Participants) | 2099 | 2132 | 4231
Age, Customized [Number; unit: participants]
  18-59 years | 706 | 734 | 1440
  60-74 years | 671 | 689 | 1360
  75+ years | 722 | 709 | 1431
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 784 | 837 | 1621
  Male | 1315 | 1295 | 2610

OUTCOME MEASURES:

1. Primary Outcome: Hospital Discharge
Description: Whether a subject was discharged alive from the hospital or alternatively died prior to discharge.
Time Frame: From time of first contact until hospital discharge, up to 90 days.
Measure: Number; unit: participants
Arm/Group | iA-CPR | M-CPR
Number analyzed (Participants) | 2094 | 2125
participants | 196 | 233

ADVERSE EVENTS:
Arm/Group | iA-CPR | M-CPR
Serious Adverse Events (participants affected / at risk) | 11/2099 | 1/2132
Other Adverse Events (participants affected / at risk) | 242/2099 | 225/2132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iA-CPR (N=2099) | M-CPR (N=2132)
CPR related injuries (Injury, poisoning and procedural complications) | 11 (11) | 1 (1) — CPR related injuries exceeding the normally expected seriousness
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iA-CPR (N=2099) | M-CPR (N=2132)
Pneumothorax (Injury, poisoning and procedural complications) | 33 (33) | 20 (20)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 159 (159) | 176 (176)
Rib Fractures (Injury, poisoning and procedural complications) | 69 (69) | 31 (31)
Subcutaneous emphysema (Injury, poisoning and procedural complications) | 21 (21) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less